CLINICAL TRIAL: NCT03708575
Title: Risk Assessment for Corneal Ectasia Following Laser in Situ Keratomileusis
Brief Title: Evaluating Risk Factors of Post-LASIK Ectasia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, HMTAbdelmoniem, principal Investigator, Assiut University
Other Study IDs: RFinCE
Record Dates: First submitted 2018-10-10; First posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Corneal Ectasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ectasia after refractive surgery is a relatively rare complication which can lead to sight-threatening complications if not detected and treated in time. It is important to continue our quest to improve our methods of identifying absolute and relative risk factors of ectasia following various keratorefractive surgical procedures.

DETAILED DESCRIPTION:
Surgical correction of refractive errors is becoming increasingly popular. In the 1990s, the excimer laser revolutionized the field of corneal refractive surgery with PRK and LASIK, refractive lenticule extraction (ReLEx) of intracorneal tissue using only a femtosecond laser, and lately ReLEx smile (SMILE). The term LASIK (Laser in situ keratomileusis) was first used in 1990 by Pallikaris, in which a microkeratome was used to cut a hinged corneal flap, followed by excimer ablation of the stromal bed and flap repositioning . LASIK is known to be a safe refractive surgical procedure, with good refractive efficacy and predictability and is associated with rapid visual recovery with minimal risk of complications.

Most of complications are flap related and include a free cap, a button hole, an incomplete cut, flap striae, interface debris, diffuse lamellar keratitis (DLK), and epithelial ingrowth. Other complications include undercorrection, overcorrection, decentered ablation, irregular ablation, and ectasia.

Corneal ectasia is a sight-threatening complication of laser refractive surgery characterized by progressive steepening and thinning of the cornea.It is defined as progressive stromal thinning and steepening of the cornea, resulting in refractive aberrations and visual deterioration. The incidence of post- LASIK ectasia is estimated to be between 0.04% and 0.6%.Corneal ectasia has been observed to occur as early as 1 week and as late as several years after LASIK.

The main purpose of assessing risk is to determine what group or groups of people present a higher chance to develop post-LASIK ectasia. The development of postoperative ectasia varies between LASIK centers and depends on the screening tools used to screen candidates, the experience and technical skill of the surgeon, and the tools used during the surgery. Risk factors for the development of post-LASIK ectasia include young age, a personal or family history of keratoconus, forme fruste keratoconus (FFKC), high myopia, low-residual stromal bed (RSB), and deep primary keratotomy resulting in a thick flap.

Although several risk factors have been identified for the likelihood of ectasia development after keratorefractive surgeries, some cases have been reported to develop in an enigmatic way, without the prescence of any of these risk factors.

ELIGIBILITY:
Inclusion Criteria:

* All subjects presented with ectasia following LASIK

Exclusion Criteria:

* Any associated ocular pathology.
* Any previous ocular surgeries other than LASIK.
* Corneal opacities.
* Ocular trauma.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: patients presented with post-LASIK corneal ectasia
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-12-10 (Estimated); Primary Completion 2019-12-10 (Estimated); Study Completion 2020-08-10 (Estimated)

PRIMARY OUTCOMES:
Post-LASIK Ectasia | 5 minutes
  Evaluating back elevation of cornea (in numbers) , corneal curvature (in diopters) , and curvature map (in diopters) using Pentacam oculizer

SECONDARY OUTCOMES:
Absolute and relative risk factors of ectasia and their cut-off values. | 5 minutes
  Degree of refraction error (in diopters) using Autorefractometer , corneal pachymetry (in micrometers) , residual stromal bed (in micrometers) , flap thickness (in micrometers) , ablation depth (in micrometers) using Pentacam oculizer , and time between LASIK and diagnosis of ectasia (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A. Mohamed, Lecturer, Study Chair — Assiut University

REFERENCES:
- [Background] Vestergaard AH. Past and present of corneal refractive surgery: a retrospective study of long-term results after photorefractive keratectomy and a prospective study of refractive lenticule extraction. Acta Ophthalmol. 2014 Mar;92 Thesis 2:1-21. doi: 10.1111/aos.12385. PMID 24636364
- [Background] Pallikaris IG, Papatzanaki ME, Siganos DS, Tsilimbaris MK. A corneal flap technique for laser in situ keratomileusis. Human studies. Arch Ophthalmol. 1991 Dec;109(12):1699-702. doi: 10.1001/archopht.1991.01080120083031. PMID 1841579
- [Background] Pallikaris IG, Papatzanaki ME, Stathi EZ, Frenschock O, Georgiadis A. Laser in situ keratomileusis. Lasers Surg Med. 1990;10(5):463-8. doi: 10.1002/lsm.1900100511. PMID 2233101
- [Background] Deitz MR, Sanders DR, Raanan MG, DeLuca M. Long-term (5- to 12-year) follow-up of metal-blade radial keratotomy procedures. Arch Ophthalmol. 1994 May;112(5):614-20. doi: 10.1001/archopht.1994.01090170058022. PMID 8185517
- [Background] dos Santos AM, Torricelli AA, Marino GK, Garcia R, Netto MV, Bechara SJ, Wilson SE. Femtosecond Laser-Assisted LASIK Flap Complications. J Refract Surg. 2016 Jan;32(1):52-9. doi: 10.3928/1081597X-20151119-01. PMID 26812715
- [Background] Sridhar MS, Rao SK, Vajpayee RB, Aasuri MK, Hannush S, Sinha R. Complications of laser-in-situ-keratomileusis. Indian J Ophthalmol. 2002 Dec;50(4):265-82. PMID 12532491
- [Background] Santhiago MR, Giacomin NT, Smadja D, Bechara SJ. Ectasia risk factors in refractive surgery. Clin Ophthalmol. 2016 Apr 20;10:713-20. doi: 10.2147/OPTH.S51313. eCollection 2016. PMID 27143849
- [Background] Randleman JB. Evaluating risk factors for ectasia: what is the goal of assessing risk? J Refract Surg. 2010 Apr;26(4):236-7. doi: 10.3928/1081597X-20100318-02. No abstract available. PMID 20415319
- [Background] Randleman JB, Woodward M, Lynn MJ, Stulting RD. Risk assessment for ectasia after corneal refractive surgery. Ophthalmology. 2008 Jan;115(1):37-50. doi: 10.1016/j.ophtha.2007.03.073. Epub 2007 Jul 12. PMID 17624434
- [Background] Chang AW, Tsang AC, Contreras JE, Huynh PD, Calvano CJ, Crnic-Rein TC, Thall EH. Corneal tissue ablation depth and the Munnerlyn formula. J Cataract Refract Surg. 2003 Jun;29(6):1204-10. doi: 10.1016/s0886-3350(02)01918-1. PMID 12842691
- [Background] Randleman JB, Russell B, Ward MA, Thompson KP, Stulting RD. Risk factors and prognosis for corneal ectasia after LASIK. Ophthalmology. 2003 Feb;110(2):267-75. doi: 10.1016/S0161-6420(02)01727-X. PMID 12578766
- [Background] Haw WW, Manche EE. Iatrogenic keratectasia after a deep primary keratotomy during laser in situ keratomileusis. Am J Ophthalmol. 2001 Dec;132(6):920-1. doi: 10.1016/s0002-9394(01)01148-5. PMID 11730659
- [Background] Giri P, Azar DT. Risk profiles of ectasia after keratorefractive surgery. Curr Opin Ophthalmol. 2017 Jul;28(4):337-342. doi: 10.1097/ICU.0000000000000383. PMID 28594648